CLINICAL TRIAL: NCT00491439
Title: Phase 1 Study of in Vivo Confocal Microscope to Evaluate the Corneal Wound Healing After Various Ocular Surgeries
Brief Title: Using in Vivo Confocal Microscope to Evaluate the Corneal Wound Healing After Various Ocular Surgeries
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Wei-Li Chen/Associate Professor, National Taiwan University Hospital
Other Study IDs: 200702038R
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2010-11

CONDITIONS: Corneal Diseases
Keywords: in vivo confocal microscopy; vitrectomy; corneal transplantation; Epi-LASIK; wound healing
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Corneal wounds after Epi-LASIK: Corneal wounds after Epi-LASIK
- penetrating keratoplasty: Corneal wound after penetrating keratoplasty
- corneal epithelial debridement: Corneal wound after pars plana vitrectioy with corneal epithelial debridement for diabetic retinopathy

SUMMARY:
Although epi-keratome laser-assisted in situ keratomileusis (Epi-LASIK), penetrating keratoplasty and pars plana vitrectomy with corneal epithelial debridement for diabetic retinopathy are surgeries commonly performed, the time-sequential, in vivo microscopic wound healing process is not fully understood. The purpose of this study is to study the healing of corneal wounds after Epi-LASIK, penetrating keratoplasty and pars plana vitrectomy with corneal epithelial debridement for diabetic retinopathy by in vivo confocal microscopy, an easily performed and non-invasive procedure. We plan to enroll 40 eyes of 40 patients in each of these three surgeries. In Epi-LASIK, slit-lamp biomicroscopy, in vivo confocal microscopy, and visual acuity are recorded before and 1, 3, and 7 days after surgery. The eyes are examined weekly in the first month and at 3 and 6 months. For penetrating keratoplasty and pars plana vitrectomy with corneal epithelial debridement, slit-lamp biomicroscopy, in vivo confocal microscopy, and visual acuity are recorded before and weekly in the first month after surgeries and at 3 and 6 months. Selected images of the corneal basal/apical surface epithelia, stromal reactions and corneal endothelial conditions by in vivo confocal microscopy are evaluated qualitatively for the cellular morphology and density.

DETAILED DESCRIPTION:
Although epi-keratome laser-assisted in situ keratomileusis (Epi-LASIK), penetrating keratoplasty and pars plana vitrectomy with corneal epithelial debridement for diabetic retinopathy are surgeries commonly performed, the time-sequential, in vivo microscopic wound healing process is not fully understood. The purpose of this study is to study the healing of corneal wounds after Epi-LASIK, penetrating keratoplasty and pars plana vitrectomy with corneal epithelial debridement for diabetic retinopathy by in vivo confocal microscopy, an easily performed and non-invasive procedure. We plan to enroll 40 eyes of 40 patients in each of these three surgeries. In Epi-LASIK, slit-lamp biomicroscopy, in vivo confocal microscopy, and visual acuity are recorded before and 1, 3, and 7 days after surgery. The eyes are examined weekly in the first month and at 3 and 6 months. For penetrating keratoplasty and pars plana vitrectomy with corneal epithelial debridement, slit-lamp biomicroscopy, in vivo confocal microscopy, and visual acuity are recorded before and weekly in the first month after surgeries and at 3 and 6 months. Selected images of the corneal basal/apical surface epithelia, stromal reactions and corneal endothelial conditions by in vivo confocal microscopy are evaluated qualitatively for the cellular morphology and density.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving various ocular surgeries
* no previous ocular surgery
* tear break up time longer than 10 seconds
* Shirmer test II larger than 5 mm
* no presurgical corneal disease confirmed by slit lamp and in vivo confocal
* no limbus defect
* proliferative retinopathy underwent vitrectomy combining corneal epithelial scrating

Exclusion Criteria:

* can not complete follow up
* ineligible for ocular surgery
* eyelid closure incomplete
* glaucoma
* corneal defect or oculoneuropathy not caused by diabetes
* severe dry eye disease
* limbus defect
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving Epi-LASIK, penetrating keratoplasty and pars plana vitrectioy with corneal epithelial debridement for diabetic retinopathy
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-04; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
cellular morphology and density | before surgery and 1, 3, and 7 days after surgeryfirst month and at 3 and 6 months

SECONDARY OUTCOMES:
corneal basal/apical surface epithelia, stromal reactions and corneal endothelial conditions | before and 1, 3, and 7 days after surgery, first month and at 3 and 6 months
visual acuity | before and 1, 3, and 7 days after surgery, first month and at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fung-Rong Hu, MD, Principal Investigator — Department of Ophthalmology, National Taiwan Universtiy Hospital
Locations (1):
- Wei-Li Chen, Taipei, Taiwan

REFERENCES:
- [Derived] Chen WL, Shen EP, Hsieh YT, Yeh PT, Wang TJ, Hu FR. Comparison of in vivo confocal microscopic findings between epi-LASIK procedures with different management of the epithelial flaps. Invest Ophthalmol Vis Sci. 2011 Jun 1;52(6):3640-7. doi: 10.1167/iovs.10-6390. PMID 21357404